CLINICAL TRIAL: NCT06445712
Title: Examining the Role of Pain in the Link Between Early Childhood Adversity and Psychopathology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202312107; UL1TR002345 (NIH)
Record Dates: First submitted 2024-05-22; First posted 2024-06-06 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Child Development
Keywords: Pain; Early Life Adversity
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain Assessment (Experimental): Children will submerge their hand in cold water and be asked to hold it in as long as possible. They will do this both alone and holding the hand of a parent (counterbalanced).
  Interventions: Behavioral: Parental Support Cold Pressor Task

INTERVENTIONS:
Behavioral: Parental Support Cold Pressor Task — Child will submerge their hand in cold water alone and holding the hand of a parent.

SUMMARY:
The goal of this study is to investigate the role of physical pain in the link between childhood adversity and later psychopathology. Children who are participating in a larger longitudinal study will be asked to submerge their hand in cold water and hold it in the cold water as long as possible. Participants will do this twice, once alone and once holding the hand of their parent, to examine the role of parental support in pain development. The study will examine self-report of pain and salivary cortisol response to pain. It is hypothesized that children who have been exposed to more adversity will experience increased pain response and increased psychopathology symptoms. It is expected that higher social support in the family will decrease this relationship.

DETAILED DESCRIPTION:
This study will initiate a program of prospective research, linking early life adversity to both pain and psychopathology symptoms in the pre-adolescent period. This study will examine these links using an existing longitudinal sample of 6.5-9.5 year-old children experiencing familial stress. The project will examine the relationship between dysregulation and pain sensitivity from the behavioral perspective, but also through HPA axis dysregulation. Finally, the project will probe parental support as a moderator on the relationship between dysregulation and pain and psychopathology symptoms. The project will use a novel adaptation of the cold pressor test to examine experimental pain sensitivity as a function of parental support by including a condition in which the child holds the hand of their parent during the task. The project will also examine the neural basis of social support through parent-child brain synchronization. Support for the proposed model may indicate that interventions that increase parental support might decrease both pain and psychopathology.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been enrolled in our ongoing CARE study

Exclusion Criteria:

* Subjects who have not participated in the CARE study

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-23 (Actual); Study Completion 2025-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for Child Brain Development, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pain Assessment
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pain Assessment
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.55 (1.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Pain Tolerance
Description: Time hand is held in cold water
Time Frame: 0-120 seconds
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Pain Assessment
Number analyzed (Participants) | 39
seconds
  Time Alone | 44.72 (35.51)
  Time Parent | 45.09 (35.91)

2. Primary Outcome: Pain Sensitivity
Description: Self-reported score on the Visual Analogue Scale for Pain. Participants use a physical sliding scale to indicate how much pain they experienced [ higher numbers are equal to more pain; (no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)]
Time Frame: 0-60 seconds after experiencing stimulus
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pain Assessment
Number analyzed (Participants) | 39
units on a scale
  VAS_Alone | 5.87 (2.79)
  VAS_Parent | 5.13 (2.67)

ADVERSE EVENTS:
Time Frame: From start of data collection on participation day to subject leaving the laboratory (approximately 1.5 to 2 hours)
Arm/Group | Pain Assessment
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT06445712/Prot_SAP_000.pdf